CLINICAL TRIAL: NCT04568733
Title: Comparison of Cardiorespiratory System Responses During Pilates Exercises and Walking
Brief Title: Cardiorespiratory Responses to a Pilates Training Session and Treadmill Walking in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-GOKAE-0133
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resting (No Intervention)
- Pilates exercise session (Experimental)
  Interventions: Behavioral: Pilates exercise session
- Treadmill walking at 3.2 kph (Active Comparator)
  Interventions: Behavioral: Treadmill walking at 3.2 kph
- Treadmill walking at 4.8 kph (Active Comparator)
  Interventions: Behavioral: Treadmill walking at 4.8 kph

INTERVENTIONS:
Behavioral: Pilates exercise session — The Pilates session will consist of warm-up exercises (e.g. breathing, arm circle, cat and camel spinal rotation etc.) and basic mat exercises (e.g. one leg stretching, double leg stretching, the hundred, saw, rolling like a ball, swimming, pelvic curl etc.). The Pilates session will be presented to the participants via pre-recorded video.
  Arms: Pilates exercise session
Behavioral: Treadmill walking at 3.2 kph — Participants will walk on a treadmill at 3.2 kph (2 mph) speed for 10 minutes.
  Arms: Treadmill walking at 3.2 kph
Behavioral: Treadmill walking at 4.8 kph — Participants will walk on a treadmill at 4.8 kph (2 mph) speed for 10 minutes.
  Arms: Treadmill walking at 4.8 kph

SUMMARY:
Low cardiorespiratory fitness is related cardiovascular and total mortality. In addition, disease risk is increased with low cardiorespiratory fitness. There is strong evidence that physical activity and cardiorespiratory fitness are associated with health variables in healthy individuals. Pilates exercises, which are the subgroups of physical activity, has become popular in recent years. Current evidence suggests that Pilates training improves body composition, respiratory muscle strength, exercise performance and quality of life. In addition to these benefits, recent evidence suggests that Pilates training can improve cardiorespiratory fitness. However, there is lack of evidence on whether practicing Pilates exercises satisfy recommendations for intensity of physical activity which improves and maintains health and cardiovascular fitness.

The primary aim of this study is to evaluate the cardiorespiratory responses during a Pilates training session, by measuring cardiorespiratory fitness through oxygen consumption and energy expenditure. The secondary aim of this study is to compare the cardiorespiratory responses during Pilates training session and treadmill walking at different speeds (3.2 kmh and 4.8 kmh).

First, resting metabolic rate will be measured. Then, the participants will be randomized to one of the two possible experimental conditions: (1) Pilates training session than treadmill walking or (2) treadmill walking than Pilates training session. Pilates session will consist of warm-up exercises (e.g. breathing, arm circle, cat and camel spinal rotation etc.) and basic mat exercises (e.g. one leg stretching, double leg stretching, the hundred, saw, rolling like a ball, swimming, pelvic curl etc.). The Pilates session will be presented to the participants via recorded video. Participants will walk on treadmill at two different speeds: 3.2 kph (2 mph) and 4.8 kph (3 mph). Participants initially will walk at pace of 3.2 kph for 10 minutes. After 30-40 minutes- rest (after returning baseline values), participants will walk on at pace of 4.8 kph for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy (not having any known chronic disease)
* Volunteer to participate in the study.

Exclusion Criteria:

* Pregnancy
* Previous disorder/surgery history that can alter physical performance in walking or Pilates session.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Oxygen Consumption (VO2) | Through basal metabolic rate assessment completion (20 minutes), through Pilates session completion (45 minutes), through treadmill walking at 3.2 kph speed completion (10 minutes), through treadmill walking at 4.8 kph speed completion (10 minutes).
  Cardiopulmonary exercise testing system will be used to oxygen consumption (L/kg/min) assessments. Oxygen consumption is an indicator of aerobic capacity. Higher scores indicate higher aerobic capacity. The mean of oxygen consumption will be recorded for resting state, Pilates session, treadmill walking at 3.2 kph speed, and treadmill walking at 4.8 kph.
Energy Expenditure | Through basal metabolic rate assessment completion (20 minutes), through Pilates session completion (45 minutes), through treadmill walking at 3.2 kph speed completion (10 minutes), through treadmill walking at 4.8 kph speed completion (10 minutes).
  A cardiopulmonary exercise testing system will be used to assess energy expenditure (kcal/min). Higher scores indicate higher energy expenditure. The mean of energy expenditure will be recorded for resting state, Pilates session, treadmill walking at 3.2 kph speed, and treadmill walking at 4.8 kph.
Metabolic Equivalent of Task (MET) | Through basal metabolic rate assessment completion (20 minutes), through Pilates session completion (45 minutes), through treadmill walking at 3.2 kph speed completion (10 minutes), through treadmill walking at 4.8 kph speed completion (10 minutes).
  Metabolic Equivalent of Task (MET) defines the expression of the intensity of physical activity. 1 MET is the rate of energy expenditure while at rest, set by convention at 3.5 mL of oxygen per kilogram per minute (mL.kg.min-1). A cardiopulmonary exercise testing system will be used to assess the MET values. Higher scores indicate higher exercise intensity. The mean of MET will be recorded for resting state, Pilates session, treadmill walking at 3.2 kph speed, and treadmill walking at 4.8 kph.

SECONDARY OUTCOMES:
Heart Rate | Through basal metabolic rate assessment completion (20 minutes), through Pilates session completion (45 minutes), through treadmill walking at 3.2 kph speed completion (10 minutes), through treadmill walking at 4.8 kph speed completion (10 minutes).
  Heart rate (beats.min-1) will be assessed using a heart rate monitor. The chest strap will be secured to participants against their skin below the sternum. Higher scores indicate higher heart rate. The mean of heart rate will be recorded for resting state, Pilates session, treadmill walking at 3.2 kph speed, and treadmill walking at 4.8 kph.
Maximum Heart Rate (%MHR) | Through basal metabolic rate assessment completion (20 minutes), through Pilates session completion (45 minutes), through treadmill walking at 3.2 kph speed completion (10 minutes), through treadmill walking at 4.8 kph speed completion (10 minutes).
  Maximum Heart Rate (%MHR) will be assessed using a heart rate monitor. Heart rate data will be multiplied by 100 and divided by the predicted maximum heart rate to determine the percentage of maximum predicted heart rate (%MHR) achieved by each individual. Higher scores indicate higher exercise intensity. The mean of %MHR will be recorded for resting state, Pilates session, treadmill walking at 3.2 kph speed, and treadmill walking at 4.8 kph.
The International Physical Activity Questionnaires (IPAQ) - short form | At baseline
  The International Physical Activity Questionnaires (IPAQ) - short form will be used to inquire about the physical activity levels of the participants. This questionnaire consists of seven questions asking participants to remind the last week's physical activity. The IPAQ-short form inquiries about the number of days and amount of the spent walking, sitting or participating in moderate (e.g., bicycling at a regular pace) and vigorous-intensity activities (e.g., fast bicycling, digging) and reports the frequency and duration of these activity. Higher scores indicate higher levels of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided